CLINICAL TRIAL: NCT05517629
Title: Face Mask Habits and COVID-19: A Cross-Sectional Study of University Students During the Third Wave in Greater Cairo
Brief Title: Face Mask Habits and COVID-19 Among University Students in Cairo
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Manar Ahmed Kamal, Principal Investigator, Benha University
Other Study IDs: FMASU R 59/2021
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Face Mask Squeeze; COVID-19; Pandemic, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- All the time: Students who wore face masks all the time when outside
  Interventions: Other: It is an observational cross-sectional study
- Most of the time: Students who wore face masks most of the time when outside
  Interventions: Other: It is an observational cross-sectional study
- Only when told to: Students who wore face masks only when they were told to when outside
  Interventions: Other: It is an observational cross-sectional study
- Not At All: Students who did not wear face masks at all when outside
  Interventions: Other: It is an observational cross-sectional study

INTERVENTIONS:
Other: It is an observational cross-sectional study — It is an observational cross-sectional study

SUMMARY:
The World Health Organization officially declared the pandemic caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) as a public health emergency. The virus can remain viable in aerosol form for approximately three hours before being inhaled. Face masks have become an essential component of the ensuing fight against coronavirus disease 2019 (COVID-19).Therefore, a multicenter cross-sectional study was conducted during the pandemic to investigate university students' face mask habits in Greater Cairo, Egypt.

DETAILED DESCRIPTION:
Study design and participants:

This cross-sectional study is going to be carried out at a time when wearing masks in public places, transportation and universities is mandatory. The questionnaire which is designed to collect the data is targeted to college students who are attending universities in Greater Cairo, Egypt. The questionnaire will be left open for a duration of 10 days to collect the required responses.

Data collection:

The data is going to be collected from a questionnaire that we created using Google forms, consisting of 33 questions. It was written in English then translated to Arabic to be understandable to as many people as possible. The survey will be sent using a snowball sampling method to the participants through various social media applications such as: Facebook, Twitter, WhatsApp, Snapchat, and Telegram. A pilot study of the questionnaire will be pre-tested on a small sample of participants to confirm the practicability and clarity of questions to check content and face validity. In addition, the reliability will be determined by calculating Cronbach alpha. Observations of the pilot study will not be included in the final analysis.

Statistical analysis:

Dichotomous data will be expressed by numbers and frequency. Continuous variables will be expressed by means and standard deviation if within the normal distribution. Range and interquartile range will be used to express continuous data within the non-normal distribution. Data will be exported to an excel sheet from Google forms and will be analyzed by an expert using IBM SPSS Statistics program.

ELIGIBILITY:
Inclusion Criteria:

* The target population was limited to individuals aged 18 to 28 years, as those individuals can provide consent and represent the undergraduate and graduate sections.
* The participants were asked about the location of their campuses to ensure that their responses were limited only to the universities in Greater Cairo.

Exclusion Criteria:

* Individuals below the age of 18 years old are not old enough to provide consent, and individuals above the age of 28 are considered postgraduate.
* To make sure that responses arrived only from Greater Cairo universities, a question asking about the location of university campus is added to exclude responses from outside the specified area which only includes the cities of Cairo, Giza, Helwan (15th of May), Shubra El Kheima, 6th of October, Sheikh Zayed City, Badr, New Cairo (including Rehab and Fifth Settlement), New Heliopolis, Obour, Shorouk, Madinaty21.

Ages: 18 Years to 28 Years | Sex: All
Age Groups: Adult
Study Population: University students who are attending universities in Greater Cairo, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 1455 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Face Mask Habits | April 20, 2021
  To evaluate participants' attitudes regarding face masks, the questions were grouped into two aspects: face mask habits (14 items) and COVID-19. Scoring Grade are four grades 1. Using face mask at all, 2. Using face mask most of time, 3. Using face mask when you are told to, and 4. Not using face mask.

CONTACTS AND LOCATIONS:
Overall Officials: Manar A Kamal, MBBCh, Principal Investigator — Benha University
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided